CLINICAL TRIAL: NCT02064569
Title: An Open Label Dose Escalation Clinical Trial to Evaluate the Safety and the Tolerability of GS010 (rAAV2/2-ND4) in Patients With Leber Hereditary Optic Neuropathy Due to Mutations in the Mitochondrial NADH Dehydrogenase 4 Gene
Brief Title: Safety Evaluation of Gene Therapy in Leber Hereditary Optic Neuropathy (LHON) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-LHON/CLIN/01
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Leber Hereditary Optic Neuropathy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GS010 (Experimental)
  Interventions: Genetic: GS010

INTERVENTIONS:
Genetic: GS010

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability profile of ascending doses of GS010 in Leber Hereditary Optic Neuropathy (LHON) patients.

ELIGIBILITY:
Inclusion Criteria:

Documented diagnosis of LHON based on a genetic test confirming the presence of the G11778A mutation in the mitochondrial ND4

Age 18 years old or older at the time of study entry (informed consent signature)

Visual acuity ≤ 1/10 of the less functional eye

Exclusion Criteria:

Any known allergy or hypersensibility to one of the product used during the trial

Contraindication to IVT surgery (anaemia Hb <8g/dl, severe cardiovascular disease, severe coagulopathy…)

Disorder of the ocular humors and of the internal retina involving visual disability

Glaucoma

Presence of other pathology whose symptoms or associated treatments might affect the retina or the optic nerve Vascular retinal occlusion

Narrow angle contra-indicating pupillary dilation

Other cause of optic neuropathy (inflammatory conditions or exposure to toxins...)

Patients presenting known mutation of other genes implicated in pathological retinal conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of local and general adverse events and Serious Adverse Events | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CATHERINE VIGNAL, MD, Principal Investigator — CIC CHNO DES QUINZE VINGTS
Locations (1):
- CIC du CHNO DES QUINZE-VINGTS, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor web site — http://www.gensight-biologics.com/